CLINICAL TRIAL: NCT00530335
Title: An Open-Label Pilot Study for Atomoxetine in Adult Subjects With Attention Deficit/Hyperactivity Disorder
Brief Title: Atomoxetine Phase 2 Study in Japanese Adult Patients With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11821; B4Z-JE-LYED (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — 40 mg/day every day (QD), by mouth (PO), for 1 week; 80 mg/day every day, by mouth, for 1 week; 105 mg/day every day, by mouth, for 2 weeks; 120 mg/day every day, by mouth, for 4 weeks
  Other Names: LY139603; Strattera

SUMMARY:
The objective is to assess overall safety and tolerability of atomoxetine in doses up to 120 mg/day in Japanese adult patients who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for ADHD

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* meet Conners' Adult ADHD Diagnostic Interview for DSM-IV™ (CAADID) diagnostic criteria for current ADHD as well as meeting criteria for a historical diagnosis of ADHD during childhood
* have a Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) score of 4 (moderate symptoms) or greater

Exclusion Criteria:

* Patients who meet DSM-IV diagnostic criteria for current major depression and also patients who have total score of more than 12 on the Hamilton Depression Rating Scale-17 items (HAMD-17) at Visit 1 and Visit 2. Patients who have both a current or past history of major depression and have received any anti-depression drug therapy within 6 months of Visit 1.
* Patients who meet DSM-IV diagnostic criteria for have a current anxiety disorder and also require anti-anxiety drug therapy except for those taking benzodiazepines analogues for anxiety which need to be limited.
* Patients who have any history of bipolar disorder (DSM-IV), any history of schizophrenia or any history of a psychotic disorder (DSM-IV) will be excluded from the study.
* Patients who have been diagnosed (DSM-IV) with a pervasive developmental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- [Result] Takahashi M, Takita Y, Goto T, Ichikawa H, Saito K, Matsumoto H, Tanaka Y. An open-label, dose-titration tolerability study of atomoxetine hydrochloride in Japanese adults with attention-deficit/hyperactivity disorder. Psychiatry Clin Neurosci. 2011 Feb;65(1):55-63. doi: 10.1111/j.1440-1819.2010.02159.x. PMID 21265936
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine: 40 mg/day every, by mouth, for 1 week; 80 mg/day every day, by mouth, for 1 week; 105 mg/day every day, by mouth, for 2 weeks; 120 mg/day every day, by mouth, for 4 weeks
Period: Overall Study
Arm/Group | Atomoxetine
Started | 45
Completed | 39
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 33.12 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 19
Region of Enrollment [Number; unit: participants]
  Japan | 45
Race/Ethnicity [Number; unit: participants]
  Japanese | 45
Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Measures severity of the patient's overall severity of attention-deficit/hyperactivity disorder (ADHD) symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 5.0 (0.8)
Conners' Adult ADHD Rating Scale-Inv:SV-J ADHD Index Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Investigator:Screening Version-Japanese. ADHD Index Subscale consisted of 12 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 36.
  units on a scale | 22.3 (5.7)
Conners' Adult ADHD Rating Scale-Inv:SV-J Hyperactive/Impulsive Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Investigator:Screening Version-Japanese. Hyperactive/Impulsive Subscale consisted of 9 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 27.
  units on a scale | 9.8 (6.2)
Conners' Adult ADHD Rating Scale-Inv:SV-J Inattentive Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Investigator:Screening Version-Japanese. Inattention subscale consisted of 9 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 27.
  units on a scale | 21.5 (3.0)
Conners' Adult ADHD Rating Scale-Inv:SV-J Total Symptoms Score [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Investigator Rating:Screening Version-Japanese . Total ADHD symptom score consisted of 18 items (sum of inattention and hyperactivity-impulsivity subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54.
  units on a scale | 31.2 (7.0)
Conners' Adult ADHD Rating Scale-S:SV-J ADHD Index Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Subject:Screening Version-Japanese. ADHD Index Subscale consisted of 12 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 36.
  units on a scale | 21.0 (6.8)
Conners' Adult ADHD Rating Scale-S:SV-J Hyperactive/Impulsive Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Subject:Screening Version-Japanese. Hyperactive/Impulsive Subscale consisted of 9 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 27.
  units on a scale | 10.1 (5.8)
Conners' Adult ADHD Rating Scale-S:SV-J Inattentive Subscale [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Subject:Screening Version-Japanese. Inattention subscale consisted of 9 items, using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 27.
  units on a scale | 19.0 (5.7)
Conners' Adult ADHD Rating Scale-S:SV-J Total Symptoms Score [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Subject:Screening Version-Japanese. Total ADHD symptom score consisted of 18 items (sum of inattention and hyperactivity-impulsivity subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54.
  units on a scale | 29.1 (9.7)
Hamilton Anxiety Rating Scale-14 Items Total Score [Mean (Standard Deviation); unit: units on a scale] — The 14-item HAMA assesses the severity of anxiety. The investigator talked to the patient about their symptoms over the previous week before the study visit. Each item was scored using a 5-point scale, i.e. 0 = absent to 4 = severe. The total score of HAMA-14 may range from 0 (normal) to 56 (severe).
  units on a scale | 6.2 (5.3)
Hamilton Depression Rating Scale-17 Items Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 4.2 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Time Frame: over 8 weeks
Population: All three participants who discontinued due to an adverse event were on atomoxetine doses of between 80 mg/day and 105 mg/day.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
participants
  Nausea | 1
  Malaise | 1
  Anorexia | 1

2. Secondary Outcome: Change From Endpoint to Baseline in Connors's Adult ADHD Rating Scale-Investigator Rated: Screening Version - Japanese Version (CAARS-Inv:SV-J)
Description: Scale=30 items divided between 3 subscales: inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items), using a 4-point scale (0=not at all/never to 3=very much/very frequently). Total ADHD symptom score consisted of 18 items (sum of inattention and hyperactivity-impulsivity subscales) with range of scores from 0 to 54.
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale
  Total ADHD Symptoms Score | -15.0 (9.0)
  Inattentive Subscale | -9.9 (6.7)
  Hyperactivity/Impulsive Subscale | -5.0 (4.6)
  ADHD Index Subscale | -9.3 (6.4)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Total ADHD Symptoms Score (endpoint - baseline)
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Inattentive Subscale scores (endpoint - baseline)
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Hyperactivity/Impulsive Subscale scores (endpoint - baseline)
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in ADHD Index Subscale scores (endpoint - baseline)

3. Secondary Outcome: Change From Endpoint to Baseline in Connors's Adult ADHD Rating Scale-Self Report: Screening Version - Japanese Version (CAARS-S:SV-J)
Description: as for outcome 2
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale
  Total ADHD Symptoms Score | -11.9 (10.6)
  Inattentive Subscale | -7.0 (7.0)
  Hyperactive/Impulsive Subscale | -4.9 (4.8)
  ADHD Index Subscale | -6.4 (6.8)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Total ADHD Symptoms Score (endpoint - baseline)
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Inattentive Subscale scores (endpoint - baseline)
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in Hyperactive/Impulsive Subscale scores (endpoint - baseline)
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value comparing difference in ADHD Index Subscale scores (endpoint - baseline)

4. Secondary Outcome: Change From Endpoint to Baseline in Clinical Global Impression-ADHD - Severity
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale | -1.2 (1.2)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Change From Endpoint to Baseline in Hamilton Depression Rating Scale - 17 Items (HAMD-17) Total Score
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale | 0.2 (4.2)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.749, t-test, 2 sided

6. Secondary Outcome: Change From Endpoint to Baseline in Hamilton Anxiety Rating Scale - 14 Items (HAMA) Total Score
Description: The 14-item HAMA assesses the severity of anxiety. The investigator talked to the patient about their symptoms over the previous week before the study visit. Each item was scored using a 5-point scale, i.e. 0 = absent to 4 = severe. The total score of HAMA-14 may range from 0 (normal) to 56 (severe).
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale | -0.1 (6.2)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.886, t-test, 2 sided

7. Secondary Outcome: Change From Endpoint to Baseline in 36-item Short-Form Health Survey (SF-36v2) Norm-based Subdomain and Summary Scores
Description: Derivation of norm-based scoring: Items re-scored to ensure choices were in consistent order and sum up converted score in each subscale; Transform subscale score; Normalize transformed subscale score (i.e. Z-score) using Japanese mean and standard deviation of SF-36v2 subscales.
  Calculate: norm-based score=Z-score*10+50 in each subscale.
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
units on a scale
  Physical Component Summary Baseline | 47.9 (9.52)
  Physical Component Summary Change from Baseline | 1.20 (9.64)
  Mental Component Summary Baseline | 44.46 (7.26)
  Mental Component Summary Change from Baseline | 0.86 (6.61)
  Physical Functioning Baseline | 54.74 (5.42)
  Physical Functioning Change from Baseline | -0.63 (4.94)
  Role-Physical Baseline | 44.04 (13.16)
  Role-Physical Change from Baseline | 2.20 (13.37)
  Bodily Pain Baseline | 49.55 (11.43)
  Bodily Pain Change from Baseline | 0.78 (10.28)
  General Health Perception Baseline | 48.30 (10.12)
  General Health Perception Change from Baseline | 0.91 (7.21)
  Vitality Baseline | 43.41 (10.22)
  Vitality Change from Baseline | 1.23 (8.73)
  Social Functioning Baseline | 43.21 (14.31)
  Social Functioning Change from Baseline | 1.17 (13.54)
  Role-Emotional Baseline | 39.09 (14.16)
  Role-Emotional Change from Baseline | 2.64 (13.54)
  Mental Health Baseline | 43.18 (10.45)
  Mental Health Change from Baseline | 1.80 (7.63)

8. Secondary Outcome: Change From Endpoint to Baseline in Stroop Color Word Test
Description: An assessment of response inhibition. Three timed tests: reading color words in black ink; reading the printed colored ink; and reading color words printed in different colored ink. There were 100 items for each of the three test categories and if they made it through the 100 words with time remaining, they would repeat the list.
Time Frame: baseline and 8 weeks
Population: All enrolled participants with Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
number of correct answers
  Word Test Baseline | 91.3 (17.9)
  Word Test Change from Baseline | 4.1 (9.2)
  Color Test Baseline | 72.8 (14.6)
  Color Test Change from Baseline | 4.9 (7.8)
  Color-Word Test Baseline | 51.7 (11.9)
  Color-Word Test Change from Baseline | 4.2 (8.8)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — P-value for comparing differences in Word Test number of correct responses (endpoint - baseline)
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for comparing differences in Color Test number of correct responses (endpoint - baseline)
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — P-value for comparing differences in Color-Word Test number of correct responses (endpoint - baseline)

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs During the Study
Description: Vital signs reported are Pulse (beats per minute [bpm]), Systolic Blood Pressure (SBP) (mmHg), and Diastolic Blood Pressure (DBP) (mmHg).
Time Frame: over 8 weeks
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
participants
  High Pulse(bpm)=Increase ≥15 to a value >120 | 0
  Low Pulse(bpm)=Decrease ≥15 to a value <50 | 0
  High SBP(mmHg)=Increase ≥20 to value at least 180 | 0
  Low SBP(mmHg)=Decrease ≥20 to value of at most 90 | 1
  High DBP(mmHg)=Increase ≥15 to value at least 105 | 0
  Low DBP(mmHg)=Decrease ≥15 to value of at most 50 | 0

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Body Weight During the Study
Description: Potentially clinically significant weight loss was defined as any decrease of at least 7%. Potentially clinically significant weight gain was defined as any increase of at least 7%.
Time Frame: over 8 weeks
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
participants
  Weight Loss=Any Decrease of at Least 7% | 4
  Weight Gain=Any Increase of at Least 7% | 0

11. Secondary Outcome: Number of Participants With Abnormal QTc Interval Based on International Conference on Harmonisation Criterion
Description: The Fridericia correction of the QT interval(QTcF) was used.
Time Frame: over 8 weeks
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
participants
  QTcF Interval of >450 milliseconds (ms) | 1
  QTcF Interval of >480 milliseconds | 0
  QTcF Interval of >500 milliseconds | 0
  QTcF Interval increase from baseline of ≥30 msec | 4
  QTcF Interval increase from baseline of ≥60 msec | 0

12. Secondary Outcome: Cytochrome P450 2D6 (CYP2D6) Phenotype Status
Description: CYP2D6 is the primary atomoxetine metabolizing enzyme. Metabolizer status was determined by focusing on the normal, decreased, and defective allele. Poor metabolizer = defective/defective. Extensive metabolizer is all except for poor metabolizer.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 45
participants
  Extensive Metabolizer | 44
  Poor Metabolizer | 1

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 45/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=45)
Palpitations (Cardiac disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 21 (24)
Stomach discomfort (Gastrointestinal disorders) | 3 (3)
Malaise (General disorders) | 6 (6)
Pyrexia (General disorders) | 3 (3)
Thirst (General disorders) | 9 (9)
Nasopharyngitis (Infections and infestations) | 16 (18)
Electrocardiogram QT prolonged (Investigations) | 3 (3)
Weight decreased (Investigations) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 11 (11)
Somnolence (Nervous system disorders) | 9 (10)
Tremor (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Middle insomnia (Psychiatric disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 4 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 6 (9)
Hot flush (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days